CLINICAL TRIAL: NCT02946645
Title: Efficiency of Neuromuscular Bite vs Physiotherapy in TMD Patients BENEFIT Study
Brief Title: Efficiency of Neuromuscular Bite vs Physiotherapy in TMD Patients
Acronym: BENEFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, PI, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16137/24.05.2016
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: TMD

STUDY DESIGN:
Intervention Model Description: Testing Bite device "A"
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Physiotherapy (Active Comparator): TMD patients will treat with orofacial physiotherapy by one expert operator according to literature
  Interventions: Procedure: Mandibular Physiotherapy
- Neuromuscular Bite (Active Comparator): TMD patients will receive an intraoral neuromuscular bite according to literature
  Interventions: Device: Neuromuscular Bite (orthotic/sub-lingual)
- Placebo (Placebo Comparator): TMD placebo group.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Neuromuscular Bite (orthotic/sub-lingual) — Bite is a device which simulates a set of properly positioned teeth
  Arms: Neuromuscular Bite
Procedure: Mandibular Physiotherapy — Mandibular Stabilisation Exercises
  1. Place knuckle of index finger between top and bottom teeth.
  2. Remove it, keeping the teeth separated one-knuckle apart.
  3. Apply gentle pressure to the to the jaw using your index finger/thumb as demonstrated in the pictures above.
  Arms: Manual Physiotherapy
Other: Placebo — No interventions.
  Arms: Placebo

SUMMARY:
Temporomandibular joint dysfunction (TMD) therapy remains an open challenge for modern dentistry. Usually physiotherapy is considered a reliable approach to treatment of TMD patients. Moreover, neuromuscular bites (orthotic) are able to reduce signs and symptoms of TMD. To our knowledge, no specific trials have been designed for the evaluation of the efficiency of physiotherapy vs neuromuscular bites in TMD patients.

The aim of this trial is to evaluate the efficiency in term of cranial muscles electromyography (sEMG), mandibular kinetic (KNG) and subjective pain scores, of orthotic vs manual physiotherapy therapy compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* myogenous TMD;
* pain duration longer than 3 months;
* presence of complete permanent dentition, with the possible exception of the third molars;
* normal occlusion.

Exclusion Criteria:

Patients were excluded from the study if they met one or more of the following criteria:

* presence of systemic or metabolic diseases;
* eye diseases or visual defects;
* history of local or general trauma;
* neurological or psychiatric disorders;
* muscular diseases;
* cervical pain;
* bruxism, as diagnosed by the presence of parafunctional facets and/or anamnesis of parafunctional tooth clenching and/or grinding;
* pregnancy;
* assumed use of anti-inflammatory, analgesic, anti-depressant, opioid, or myorelaxant - - drugs;
* smoking;
* fixed or removable prostheses;
* fixed restorations that affected the occlusal surfaces;
* and either previous or concurrent orthodontic or orthognathic treatment. For comparison with previous literature, the diagnosis of myofascial-type TMD was provided after clinical examination by a trained clinician according to group 1a and 1b of the Research Diagnostic Criteria for TMD (RDC/TMD), in a blinded manner

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Surface electromiography of cranial muscles (sEMG) | Average of 1 year
  Evaluation of surface electromiography of cranial muscles (expressed in microvolts)
Mandibular kinesiography (KNG) | Average of 1 year
  Evaluation of mandibular kinetics (expressed in millimeters/seconds)

SECONDARY OUTCOMES:
Pain scale | 15 days
  Evaluation of subjective pain perception by Visual Analog Scale (expressed in unit)

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic, University of L'Aquila, St. Salvatore Hospital,, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Toledo EG Jr, Silva DP, de Toledo JA, Salgado IO. The interrelationship between dentistry and physiotherapy in the treatment of temporomandibular disorders. J Contemp Dent Pract. 2012 Sep 1;13(5):579-83. PMID 23250156
- [Background] List T, Axelsson S. Management of TMD: evidence from systematic reviews and meta-analyses. J Oral Rehabil. 2010 May;37(6):430-51. doi: 10.1111/j.1365-2842.2010.02089.x. Epub 2010 Apr 20. PMID 20438615
- [Background] Molin C. From bite to mind: TMD--a personal and literature review. Int J Prosthodont. 1999 May-Jun;12(3):279-88. PMID 10635197
- [Background] Michelotti A, de Wijer A, Steenks M, Farella M. Home-exercise regimes for the management of non-specific temporomandibular disorders. J Oral Rehabil. 2005 Nov;32(11):779-85. doi: 10.1111/j.1365-2842.2005.01513.x. PMID 16202040
- [Background] Capellini VK, de Souza GS, de Faria CR. Massage therapy in the management of myogenic TMD: a pilot study. J Appl Oral Sci. 2006 Jan;14(1):21-6. doi: 10.1590/s1678-77572006000100005. PMID 19089025
- [Background] Ash MM Jr, Ramfjord SP. Reflections on the Michigan splint and other intraocclusal devices. J Mich Dent Assoc. 1998 Oct;80(8):32-5, 41-6. PMID 9863432
- [Background] Yamashita A, Kondo Y, Yamashita J. Thirty-year follow-up of a TMD case treated based on the neuromuscular concept. Cranio. 2014 Jul;32(3):224-34. doi: 10.1179/0886963413Z.00000000020. Epub 2014 Jan 24. PMID 25000166
- [Background] Di Fabio RP. Physical therapy for patients with TMD: a descriptive study of treatment, disability, and health status. J Orofac Pain. 1998 Spring;12(2):124-35. PMID 9656890
- [Background] Starnes LO. A bite orthotic for the resting period between two phases of treatment. J Clin Orthod. 2002 Feb;36(2):92-4. No abstract available. PMID 11902010
- [Background] Heit T. Neuromuscular orthotics in the treatment of craniomandibular dysfunction and the effects on patients with multiple sclerosis: a pilot study. Cranio. 2011 Jan;29(1):57-70. doi: 10.1179/crn.2011.009. PMID 21370770
- [Background] Cooper BC, Kleinberg I. Establishment of a temporomandibular physiological state with neuromuscular orthosis treatment affects reduction of TMD symptoms in 313 patients. Cranio. 2008 Apr;26(2):104-17. doi: 10.1179/crn.2008.015. PMID 18468270
- [Result] Pietropaoli D, Cooper BC, Ortu E, Monaco A; I.A.P.N.O.R.. A Device Improves Signs and Symptoms of TMD. Pain Res Manag. 2019 May 6;2019:5646143. doi: 10.1155/2019/5646143. eCollection 2019. PMID 31198477